CLINICAL TRIAL: NCT01208324
Title: Interaction of Estrogen and Serotonin in Modulating Brain Activation in Menopause
Brief Title: Estrogen and Serotonin on Changing Brain Chemistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 809690; P50MH099910 (NIH)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Menopause
Keywords: Cognitive difficulties; memory impairment; mood changes; brain activation
MeSH Terms: conditions — Memory Disorders | interventions — Estradiol; Amino Acids; Isoleucine; Leucine; Lysine; Methionine; Phenylalanine; Threonine; Valine; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Estrogen patch (Active Comparator): Vivelle Dot® 0.10 - 0.15 mg/day for 8 weeks
  Interventions: Drug: estrogen patch
- Amino Acids (Active Comparator): L-Isoleucine (4.2 g), L-Leucine (6.6 g), L-Lysine (4.8 g), L-Methionine (1.5 g), L-Phenylalanine (6.6 g), L-Threonine (3.0 g), L-Valine (4.8 g)
  Interventions: Drug: Amino acids; Drug: Placebo pills
- Placebo Patch (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Patch
- Placebo pills (Placebo Comparator): 31.5 g of lactose or microcellulose
  Interventions: Drug: Placebo pills

INTERVENTIONS:
Drug: estrogen patch — 150 subjects will be enrolled in a double blind placebo controlled study where they will be randomized to receive either treatment with 17β-estradiol (Vivelle Dot® 0.10 - 0.15 mg/day) or a look-alike placebo patch for a total of approximately 8 weeks. There will be four fMRI test sequences: two test sequences one week apart prior to estrogen treatment (ET) or placebo treatment (PT), and two sequences one week apart following approximately 6-weeks of double-blind ET or PT. During each test day, all subjects will have their blood drawn at specific time intervals and undergo a battery of cognitive testing.While on the ET or PT treatment, all subjects will be instructed to change the patch every 3.5 days.
  Other Names: Vivelle-Dot®
  Arms: Estrogen patch
Drug: Amino acids — 31.5 mg of amino acids or 31.5 mg of lactose will be administered to subjects on each of their 4 test days. On 2 of the test days subjects will receive the active pills (amino acids) and on the other 2 test days subjects will receive the placebo pills (lactose).
  Other Names: L-Isoleucine; L-Leucine; L-Lysine; L-Methionine; L-Phenylalanine; L-Threonine; L-Valine
  Arms: Amino Acids
Drug: Placebo Patch — placebo
  Other Names: Placebo
  Arms: Placebo Patch
Drug: Placebo pills — There are 4 test days in this study. Each test day will involve the ingestion of 70 capsules. During one of each pair of tests, the 70 capsules will contain 31.5 g of lactose (sham depletion), while during the other test they will contain a total of 31.5 g of amino acids.
  Other Names: lactose
  Arms: Amino Acids; Placebo pills

SUMMARY:
The aim of this study is to examine the effects of estrogen and serotonin on cognition, emotional processing, and brain activation. The investigators will study the effects of acute tryptophan (TRP) depletion on cognition and mood in healthy menopausal women before and after estrogen replacement treatment (ERT). Using functional magnetic resonance imaging (fMRI), the investigators will identify differences in brain activation during memory tasks with and without TRP depletion and before and after estrogen therapy in order to determine which brain regions and cognitive functions are affected by each manipulation.

DETAILED DESCRIPTION:
The overarching purpose of this study is to further our understanding of the individual and interactive effects of the hormone estrogen and the neurotransmitter serotonin on certain aspects of cognition and brain activation in menopausal women ages 48 to 60 years. Women will undergo cognitive testing and fMRI sessions both before and after 6 weeks of either estrogen or placebo administration. We will recruit women who are across the first 10 years since their last menstrual period so that the investigators can gather information regarding the potential impact of time since menopause on our outcomes of interest. We anticipate that findings from this study will help scientist and clinicians to refine their use of estrogen therapy in menopausal women. In addition, should the role of serotonin be of utmost importance for maintenance of healthy cognition, these data aid future drug development to preserve health cognition and/or to treat dementias in which serotonin is an important factor. This proposal is both novel and timely as results from this study are likely to provide information critical to the on-going discussion regarding the risks and benefits of ET use in menopausal women.

ELIGIBILITY:
Key Inclusion Criteria:

Women ages 48 to 60 (at the time of enrollment) will be eligible for this study if they:

1. Have no history of major depressive disorder, generalized anxiety disorder, and or panic disorder within the last three years according to the Structured Clinical Interview for DSM-IV (Diagnostic and Statistical Manual) Axis I Disorders (SCID-NP) (First et al., 1995), or a history of major depressive disorder, generalized anxiety disorder, and or panic disorder greater than 3 years ago, but now resolved according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP) (First et al., 1995);
2. Have no substance abuse disorders (this includes alcohol, prescription, and illicit substances) within the last three years according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP) (First et al., 1995);
3. Subject has history of substance abuse disorders (this includes alcohol, prescription, and illicit substances) >3 years ago but the period of abuse did not last more than 5 years according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP) (First et al., 1995);
4. No first-degree relative (excluding children) with a known psychotic disorder or bi-polar disorder per patient report. Psychotic disorders include schizophrenia, schizoaffective disorder, psychotic disorder;
5. Have not taken hormonal contraceptives, ET (estrogen therapy) or HT (hormone therapy) for at least 3 months as per self-report;
6. Are within 10 years and 11 months of LMP (last menstrual period) as per self-report;
7. Have a follicular stimulating hormone level (FSH) of >30 IU/ml as per hormone testing results; women with an FSH below 30 will have the option to undergo an additional blood draw between 3-9 months following the initial blood draw (see note 2 below);
8. Are able to give written informed consent;
9. Provide written documentation of having had a normal mammogram and a PAP smear (Papanicolaou test) within the recommended timeframe as defined by the American College of Obstetricians and Gynecologists (ACOG) - please visit their website for current recommendations;
10. Must have clear urine toxicology screen upon recruitment;
11. Are fluent in written and spoken English;
12. Are right-handed.

Key Exclusion Criteria

1. Currently smoking more than 10 cigarettes/day by self report;
2. History of clinical CVD (cardiovascular disease) including myocardial infarction, angina, or congestive heart failure;
3. History of thromboembolic disease (deep vein thrombosis or pulmonary embolus);
4. History of untreated (no cholecystectomy) gallbladder disease as per self-report during PE;
5. History of triglyceridemia by subject report;
6. Undiagnosed vaginal bleeding as per self-report;
7. History of estrogen responsive cancers as per self-report;
8. Known hypercoagulable state (thrombophilias) as per self-report;
9. Severe lactose intolerance (sham depletion requires lactose/microcellulose administration; mild to moderate lactose intolerance is acceptable); Dr. Epperson will make the final decision whether an individual's lactose intolerance is severe enough to require exclusion;
10. Use of estrogen- or progestin-containing medication or phytoestrogen containing supplements (e.g. soy concentrates or extracts) within 3 months of participation as per self-report; foods containing soy (e.g. tofu, soy milk) will be permissible; estrogen-based localized treatments such as creams and vaginal inserts will be permissible, so long as said treatments do not effect systemic estrogen levels (women using localized treatments must have estrogen levels similar to other women in the study of their age and menopause status). PI will have final decision about enrollment (see note 3 below);
11. Have a Mini Mental Status Score of < 25;
12. Hamilton Depression Score > 14;
13. As per self-report, have taken a psychotropic medication within the previous month, with the exception of sleeping aids if the participant is willing to forgo use during study participation;
14. Have a metallic implant as per self-report;
15. Are claustrophobic as per self-report;
16. Are pregnant (pertains to peri-menopausal women only).

Note 1: In the case of participants with full or partial hysterectomy, timing of final menstrual period will be determined by Dr. Epperson (the study PI) or one of the study MDs. In cases in which final menstrual period cannot be established, subjects will be excluded from the study.

Note 2: Women who undergo the repeat FSH blood test will be enrolled if their levels are > 30. Women will not be required to repeat all admission procedures unless they report experiencing a life event which would impact their mental or physical health and well-being. The PI will make the final determination regarding what, if any, screening procedures need to be repeated.

Note 3: Women on localized estrogen treatments who show elevated systemic estrogen levels will not be enrolled. Instead, they will need to discontinue use for 1 month and then have their estrogen levels retested with an additional blood draw. PI will have the final decision regarding eligibility.

Ages: 48 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Neill Epperson, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Center for Women's Behavioral Wellness, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epperson CN, Amin Z, Naftolin F, Cappiello A, Czarkowski KA, Stiklus S, Anderson GM, Krystal JH. The resistance to depressive relapse in menopausal women undergoing tryptophan depletion: preliminary findings. J Psychopharmacol. 2007 Jun;21(4):414-20. doi: 10.1177/0269881106067330. Epub 2006 Aug 4. PMID 16891341
- [Background] Amin Z, Gueorguieva R, Cappiello A, Czarkowski KA, Stiklus S, Anderson GM, Naftolin F, Epperson CN. Estradiol and tryptophan depletion interact to modulate cognition in menopausal women. Neuropsychopharmacology. 2006 Nov;31(11):2489-97. doi: 10.1038/sj.npp.1301114. Epub 2006 Jun 7. PMID 16760926
- [Background] Amin Z, Epperson CN, Constable RT, Canli T. Effects of estrogen variation on neural correlates of emotional response inhibition. Neuroimage. 2006 Aug 1;32(1):457-64. doi: 10.1016/j.neuroimage.2006.03.013. Epub 2006 Apr 27. PMID 16644236
- [Background] Amin Z, Canli T, Epperson CN. Effect of estrogen-serotonin interactions on mood and cognition. Behav Cogn Neurosci Rev. 2005 Mar;4(1):43-58. doi: 10.1177/1534582305277152. PMID 15886402
- [Background] Kugaya A, Epperson CN, Zoghbi S, van Dyck CH, Hou Y, Fujita M, Staley JK, Garg PK, Seibyl JP, Innis RB. Increase in prefrontal cortex serotonin 2A receptors following estrogen treatment in postmenopausal women. Am J Psychiatry. 2003 Aug;160(8):1522-4. doi: 10.1176/appi.ajp.160.8.1522. PMID 12900319
- See also: Program Website — http://www.med.upenn.edu/womenswellness/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants included in the Placebo Patch/ Active then Sham group completed Test Day 1, but did not receive a patch.
  1 participant included in the Placebo Patch/ Sham then Active group completed Test Day 1, but did not receive a patch.
Groups:
- Active Patch: Active Tryptophan, Then Sham Tryptophan: Participants assigned to receive the Active ET patch, and sequence of active tryptophan followed by sham tryptophan. There will be four successful* TRP depletion test sequences: two test sequences one week apart prior to randomization to ET or PT, and two sequences one week apart following approximately 6-weeks of double-blind ET or PT. Each TRP depletion test day will involve ingestion of 70 capsules. During one of each pair of tests, the 70 capsules will contain 31.5 g of lactose (sham depletion; for participants who are not lactose intolerant) or 31.5 g of microcellulose (sham depletion; for participants who have mild to moderate lactose intolerance), while during the other test they will contain a total of 31.5 g of amino acids, but no tryptophan.
- Active Patch: Sham Tryptophan, Then Active Tryptophan: Participants assigned to receive the Active ET patch, and sequence of sham tryptophan followed by active tryptophan. There will be four successful* TRP depletion test sequences: two test sequences one week apart prior to ET or PT, and two sequences one week apart following approximately 6-weeks of double-blind ET or PT. Each TRP depletion test day will involve ingestion of 70 capsules. During one of each pair of tests, the 70 capsules will contain 31.5 g of lactose (sham depletion; for participants who are not lactose intolerant) or 31.5 g of microcellulose (sham depletion; for participants who have mild to moderate lactose intolerance), while during the other test they will contain a total of 31.5 g of amino acids, but no tryptophan.
- Sham Patch: Active Tryptophan, Then Sham Tryptophan: Participants assigned to receive the Sham patch, and sequence of active tryptophan followed by sham tryptophan. There will be four successful* TRP depletion test sequences: two test sequences one week apart prior to randomization to ET or PT, and two sequences one week apart following approximately 6-weeks of double-blind ET or PT. Each TRP depletion test day will involve ingestion of 70 capsules. During one of each pair of tests, the 70 capsules will contain 31.5 g of lactose (sham depletion; for participants who are not lactose intolerant) or 31.5 g of microcellulose (sham depletion; for participants who have mild to moderate lactose intolerance), while during the other test they will contain a total of 31.5 g of amino acids, but no tryptophan.
- Sham Patch: Sham Tryptophan, Then Active Tryptophan: Participants assigned to receive the Sham ET patch, and sequence of sham tryptophan followed by active tryptophan. There will be four successful* TRP depletion test sequences: two test sequences one week apart prior to randomization to ET or PT, and two sequences one week apart following approximately 6-weeks of double-blind ET or PT. Each TRP depletion test day will involve ingestion of 70 capsules. During one of each pair of tests, the 70 capsules will contain 31.5 g of lactose (sham depletion; for participants who are not lactose intolerant) or 31.5 g of microcellulose (sham depletion; for participants who have mild to moderate lactose intolerance), while during the other test they will contain a total of 31.5 g of amino acids, but no tryptophan.
Period: Pre-randomization of Patch
Arm/Group | Active Patch: Active Tryptophan, Then Sham Tryptophan | Active Patch: Sham Tryptophan, Then Active Tryptophan | Sham Patch: Active Tryptophan, Then Sham Tryptophan | Sham Patch: Sham Tryptophan, Then Active Tryptophan
Started | 14 | 15 | 10 | 8
Test Day 1 (1 Sham Patch: Sham Tryptophan, then Active Tryptophan participant did not comp) | 14 | 15 | 10 | 8
Test Day 2 | 14 | 15 | 8 | 5
Completed (Five participants did not make it to Test Day 2) | 14 | 15 | 8 | 5
Not Completed | 0 | 0 | 2 | 3
Period: Post-randomization of Patch
Arm/Group | Active Patch: Active Tryptophan, Then Sham Tryptophan | Active Patch: Sham Tryptophan, Then Active Tryptophan | Sham Patch: Active Tryptophan, Then Sham Tryptophan | Sham Patch: Sham Tryptophan, Then Active Tryptophan
Started (One participant withdrew post Test Day 2) | 14 | 15 | 8 | 5
Test Day 3 | 13 | 15 | 8 | 5
Test Day 4 | 13 | 15 | 8 | 5
Completed | 13 | 15 | 8 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The participants that were analyzed completed all 4 test days. The study team was not permitted to collect or use the information collected from the 6 participants who did not complete up to test day 4, and so those participants are excluded from the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Patch: Active Tryptophan, Then Sham Tryptophan | Active Patch: Sham Tryptophan, Then Active Tryptophan | Sham Patch: Active Tryptophan, Then Sham Tryptophan | Sham Patch: Sham Tryptophan, Then Active Tryptophan | Total
Number analyzed (Participants) | 13 | 15 | 8 | 5 | 41
Age, Continuous [Mean (Full Range); unit: years] — Women ages 48-60
  years | 55.15 [49.2 to 60] | 55.69 [49.2 to 59.3] | 54.94 [48.3 to 59.9] | 54.16 [49 to 60.7] | 55.18 [48.3 to 60.7]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 13 | 15 | 8 | 5 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 0 | 6
  White | 9 | 13 | 6 | 4 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Adverse Childhood Experiences (ACE) Questionaire [Count of Participants; unit: Participants] — The ACE is used to assess history of emotional, physical, or sexual abuse, childhood neglect, and household dysfunction. The number of exposures was summed to create the ACE score (range: 0-10). Subjects with an ACE score ⩾2 were considered 'high ACE' while subjects with ACE score of < 2 were considered 'low ACE'. A threshold of 2 was used to define the high ACE group based on studies of depression prevalence in later life that demonstrate increased susceptibility at this level of exposure.
  Participants
    High ACE | 5 | 7 | 4 | 0 | 16
    Low ACE | 8 | 8 | 4 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in BOLD Signal
Description: To replicate and extend our previous behavioral findings of an interaction between estrogen therapy (ET) and tryptophan depletion on verbal memory in a group of early menopausal women randomized to receive ET. Blood-oxygen-level dependent or BOLD signal is the outcome of BOLD imaging, which is a technique used in functional MRI. BOLD signal reflects changes in regional cerebral blood flow which delineate regional activity. A positive BOLD signal marks an increase in regional blood flow, while a negative BOLD signal marks a decrease in regional blood flow. A positive percent change means that between scans the BOLD signal i.e. blood flow in that region has increased, a negative percent change means that the BOLD signal has decreased between scans.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of BOLD signal changes
Groups:
- High Ace: Participants with an adverse childhood experience (ACE) score greater than or equal to 2.
- Low Ace: Participants with an adverse childhood experience (ACE) score less than 2.
Arm/Group | High Ace | Low Ace
Number analyzed (Participants) | 16 | 24
percentage of BOLD signal changes | -.43 [-.65 to -.22] | .20 [-.16 to .21]

2. Secondary Outcome: Evaluate the Changes in Verbal Working Memory Mediated Through the Dorsolateral Prefrontal Cortex.
Description: To evaluate the extent to which effects of ET (estrogen therapy) and TRP-D on verbal working memory are mediated through the dorsolateral prefrontal cortex.
Time Frame: 8 weeks
Population: This outcome measure was not assessed. No participants were analyzed and no data was collected.
Arm/Group | High ACE | Low ACE
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was at each test day visit, of which there were 4 and over the course of the 10-week patch treatment (either Estradiol or placebo).
Arm/Group | Active Patch: Active Tryptophan, Then Sham Tryptophan | Active Patch: Sham Tryptophan, Then Active Tryptophan | Sham Patch: Active Tryptophan, Then Sham Tryptophan | Sham Patch: Sham Tryptophan, Then Active Tryptophan
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT01208324/Prot_SAP_000.pdf